CLINICAL TRIAL: NCT02828605
Title: Virtual Interactive Platform (VIP) Transplant Research Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1607018023
Record Dates: First submitted 2016-07-07; First posted 2016-07-11 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Transplant Patients
MeSH Terms: interventions — Transplantation

ARMS (2):
- Control Group (No Intervention): Only receive surveys.
- Experimental Group (Experimental): Receive VIP Transplant App and surveys.
  Interventions: Device: Virtual Interactive Platform (VIP) Transplant

INTERVENTIONS:
Device: Virtual Interactive Platform (VIP) Transplant
  Arms: Experimental Group

SUMMARY:
The purpose of this study is to test a tablet-based application called VIP Transplant, devised to improve the recovery experience of patients that have recently had organ transplant surgery. The study will consist of two non-randomized arms: the first arm will consist of usual care and the second will be using the newly developed app for 21 days to replace their in-person visits. Using questionnaires and in-app usage metrics, the research team will track whether patients have a better medical outcome, greater patient satisfaction with care, and greater compliance rates as compared to patients who do not use VIP Transplant to manage their care.

DETAILED DESCRIPTION:
An organ transplant requires a large time and financial investment for both the patient and provider over the course of a lifetime of follow-up visits and lifestyle monitoring. Patients return to the clinic 2-3 times a week for the first three months after surgery, and then visit the clinic twice a month with labs once a week 91-210 days post surgery. Check-ins for patients without complications occur 1-2 times a year, and these re-evaluations require patients to take time off work and travel to the transplant center often 2 hours away. Dr. David Mulligan, Chief of Transplant at Yale wanted to help patients reduce the time and cost associated with their regular checkups after surgery. Thus, we created VIP Transplant. The Virtual Interactive Platform allows patients to have a secure videoconference with their provider in order to eliminate the need for recurring travel and waiting in congested clinics for a short appointment. It will save patient time and cost to travel to the clinic. The application is integrated into the provider network in order to have a system that supports seamless communication between the patient and provider capabilities.

Research plan:

Dr. Mulligan will contact 8 of his patients who are willing to participate in the study. 4 of the patients will be assigned to the control group and the other 4 will be assigned to the experimental group.

Control group:

On day 1 after their surgery, patient will be asked to fill out a survey on their transplant care. On day 21, patient will be asked to fill out the same survey. The surgeon will be asked to take a survey to evaluate their each patient's progress.

Experimental group:

When the 4 patients attend orientation, patient will each be given the iPad with the VIP Transplant app and shown how to use the app. Patient will then be asked to fill out the survey on day 1 after their surgery and then asked to use VIP Transplant for their transplant care in the following days. Patient will then be asked to fill out the survey again on day 21, at the end of the study. The surgeon will be asked to take a survey to evaluate each of their patient's progress.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Familiarity with English
* Familiarity with iPad usage/technologically adept

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Time to travel from home to Yale New Haven Hospital | 30 days
  Questionnaire, Scales of 1 to 10
Cost to travel from home to Yale New Haven Hospital | 30 days
  Questionnaire, Scales of 1 to 10
Patient Satisfaction with Care | 30 days
  Questionnaire, Scales of 1 to 10
Physician Satisfaction with Care | 30 days
  Questionnaire, Scales of 1 to 10